CLINICAL TRIAL: NCT03660709
Title: A RCT Evaluating the Efficacy of Enhanced and Standard Versions of HIV Testing and Counselling Among Men Who Have Sex With Men in Hong Kong
Brief Title: Comparing the Efficacy of Enhanced and Standard HTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MSS249R
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Behavior, Sex
Keywords: Unprotected anal intercourse; HIV retesting; Risk perception
MeSH Terms: conditions — Sexual Behavior | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): enhanced version of HIV testing and counseling
  Interventions: Behavioral: Intervention
- Control (Active Comparator): standard-of-care HIV testing and counseling
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Intervention — 1. Standard-of-care HIV testing and counseling
  2. Watch a video clip while waiting for the HIV testing result on a tablet.
  3. Receive a pamphlet and post-test counselling promoting HIV retesting.
  4. Receive the e-health HIV risk calculator through e-mail, SMS or social media means 3 and 5 months afterwards.
  5. Receive brief e-health reminder for retesting at Month 3 and 5.
  Arms: Intervention
Behavioral: Control — Standard-of-care HIV testing and counseling
  Arms: Control

SUMMARY:
Objective The objectives of the study are to evaluate the relative efficacy of an enhanced version of HIV testing and counselling (EHTC) versus standard-of-care HIV testing and counselling (SHTC) in reducing sexual risk behaviours, increasing retesting rate and risk perception among men who have sex with men (MSM) in Hong Kong.

Participants Inclusion criteria are: 1) men of age 18 years or above using HTC services at AIDS Concern, 2) anal intercourse with at least one man in the last six months, 3) able to read and comprehend Cantonese, 4) willingness to provide contact information and to complete a simple follow up evaluation at Month 6, and 5) no intention to leave Hong Kong for one month consecutively within the next six months. Those self-reported or tested to be HIV positive will be excluded from the study.

Design A parallel-group and non-blinded randomized controlled trial (RCT) will be conducted. A total of 430 participants will be randomly allocated into the intervention group receiving EHTC (n=215) and the control group receiving SHTC (n=215). Evaluation will be performed six months afterwards.

Outcomes Primary outcomes are: 1) Prevalence of unprotected anal intercourse with any and specific types of male partners during the 6-month follow up period; 2) uptake of any type of HIV antibody testing within the 6-month follow-up period, and 3) HIV risk perception.

DETAILED DESCRIPTION:
Aim To evaluate the relative efficacy of an enhanced version of HIV testing and counselling (EHTC) that combines a component proven effective and new components involving e-health and HIV risk self-assessment versus standard-of-care HIV testing and counselling (SHTC) in reducing sexual risk behaviours, and increasing HIV retesting rate and risk perception among men who have sex with men (MSM) in Hong Kong.

Objectives To compare outcomes obtained from the intervention group (EHTC) and the control group (SHTC) at Month 6, including: 1) prevalence of unprotected anal intercourse with any type and specific types of male sex partners (regular and non-regular partners) in the last six months, 2) prevalence of having taken up any type of HIV antibody testing within the 6-month follow-up period, and 3) level of HIV risk perception.

Study design A parallel-group and non-blinded randomized controlled trial (RCT) will be conducted. A total of 430 participants will be randomly allocated into the intervention group receiving EHTC (n=215) and the control group receiving standard-of-care HTC (SHTC; n=215). Evaluation will be performed six month afterwards.

Recruitment procedures Users of AIDS Concern's HTC service will be approached by staff of AIDS Concern. They will brief the participants about the detail of the study and invite them to participate. Prospective participants who are interested in joining the study will be screened for their eligibility. Guarantees will be made on anonymity, right to quit at any time and that refusal will not affect their chance in using any services. Verbal instead of written informed consent will be obtained due to maintaining anonymity but the fieldworkers will sign a form pledging that the participants have been fully informed about the study.

Baseline survey and randomization Participants will complete a self-administered baseline questionnaire on site. Participants are randomized 1:1 into the intervention group and the control group. Staff of the NGO will draw one of the sealed opaque envelops to randomly allocate participants into the intervention and the control groups. Random numbers will be generated by a computer. Block randomization with block size of eight will be used.

Pre-test counselling and rapid testing All consented participants in both groups will receive the same standard-of-care pre-testing counselling, which has currently been provided by the NGO staff. It takes about five minutes to complete; it covers knowledge on HIV prevention, risk assessment, and explanation of the procedure and benefits of HTC. A rapid HIV antibody test (finger prick) will then be performed. Testing results will be known in about 15 minutes.

The control group Participants that are allocated to the control group will receive the standard-of-care HTC, which includes the previous pre-testing counselling procedures. In the post-testing counselling, participants will be explained about the negative HIV testing result (e.g. window period for screening). They will also be reminded about risk of HIV transmission, and be facilitated to set up specific goals for consistent condom use. The standard-of-care post-testing counselling lasts for about 15 minutes.

The intervention group In addition to the steps received by members of the control group, the intervention group will be exposed to four additional intervention components.

1. A video clip While waiting for the HIV testing result, participants in the intervention group will watch a 10-minute video clip presenting the story of a gay man contracting sexually transmitted diseases in Hong Kong on a tablet.
2. A pamphlet and post-test counselling promoting HIV retesting During the standard post-test counselling, the NGO staff will perform additional brief discussions about the importance of HIV retesting. A pamphlet promoting HIV retesting in the future six months will be prepared by this study and be distributed to participants after they have completed viewing the video.
3. The e-health HIV risk calculator Through e-mail, SMS or social media means, participants will be suggested 3 and 5 months after receiving the EHTC to make a self-assessment of one's own HIV-related risk through an online personalized HIV risk self-assessment.
4. Brief e-health reminder for retesting Brief SMS or social media messages will be sent to participants at Month 3 and 5.

Follow up evaluation Participants of both the intervention and control groups will be followed up six months after receiving the HTC.

Statistical analysis Intention-to-treat analysis will be conducted. Between-group (intervention versus control) baseline differences in the frequency distributions of potential confounders will be compared by using chi-square test, t-test, Mann-Whitney test or other statistics. The absolute and relative risks and number needed to treat (and their 95% confidence intervals) for the binary primary outcomes comparing the two groups at Months 6 will be derived. Adjusted comparisons between the intervention and control groups will be made for all binary outcomes, adjusting for any potential confounders showing p<.2 in the between-group baseline comparisons (if any), using modified Poisson regression with robust sandwich variance estimation. SPSS 18.0 will be used for data analysis; p<.05 (2-sided) will be taken as statistically significant. The research team is very experienced in performing data analysis.

Sample size planning Assuming the prevalence of UAI with any male partners in the last six months is 40% in the control group when measured at Month 6, a sample size of 152 per group allows us to detect a smallest between-group difference of UAI of 15% (power=0.8, alpha=0.05), taking into an expected 30% loss of follow up at Month 6. A target sample size of about 215 per group is required. The actual sample size will be 430 (215 for the intervention group and 215 for the control group).

ELIGIBILITY:
Inclusion Criteria:

* men of age 18 years or above taking up HIV testing and counselling (HTC) at a collaborative non-governmental organization (NGO),
* anal intercourse with at least one man in the last six months
* able to read and comprehend Cantonese
* willingness to provide contact information and to complete a simple follow up evaluation at Month 6
* no intention to leave Hong Kong for one month consecutively within the next six months.

Exclusion Criteria:

* self-reported or tested to be HIV positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Take up any type of HIV antibody testing | six months
  Uptake of any type of HIV antibody testing within the follow-up period will be assessed at Month 6 telephone follow-up evaluation

SECONDARY OUTCOMES:
Unprotected anal intercourse with any and specific types of male partners | six months
  Prevalence of unprotected anal intercourse with any and specific types of male partners will be recorded at Month 6 telephone follow-up evaluation
Risk perception | six months
  Perceived risk of HIV infection will be assessed at Month 6 telephone follow-up evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No